CLINICAL TRIAL: NCT01241123
Title: The Influence of Ambulation on the Return of Bowel Function After Colorectal Surgery: Traditional Care Versus Early Mobilization Protocol
Brief Title: The Influence of Ambulation on the Return of Bowel Function After Colorectal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI retired and no recruitment occurred
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP# 10-0061
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Return of Bowel Function After Colon Surgery
Keywords: return of bowel function, post-operative, colon surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Ambulation regimen (Placebo Comparator): All patients will receive pedometers to record the total amount of ambulation. These patients will ambulate without limitations or goals. Most surgeons request that post-operative patients ambulate at least 2 to 3 times a day.
  Interventions: Drug: Sitz-Markers; Radiation: Daily abdominal x-rays; Device: pedometers
- Walkers (Active Comparator): All patients will receive pedometers to record the total amount of ambulation. Patients in the experimental group will have assigned nursing staff assisting in ambulation in these patients at least three times a day.
  Interventions: Procedure: Ambulation regimen; Drug: Sitz-Markers; Radiation: Daily abdominal x-rays; Device: pedometers

INTERVENTIONS:
Procedure: Ambulation regimen — Assistance and encouragement for at least ambulation 3 times a day
  Arms: Walkers
Drug: Sitz-Markers — radiopaque markers to subjectively follow the return of bowel function
Radiation: Daily abdominal x-rays — daily abdominal x-rays for 7 days - to follow the radiopaque markers
Device: pedometers — to record the amount of ambulation

SUMMARY:
"Fast-track" or "enhanced recovery" programs, which are the new standardized accelerated clinical pathways for post-operative care for colorectal surgeries, have three goals: to 1) quicken the return of bowel function (as evidenced by passage of flatus and stool), 2) decrease the length of hospital stays, and 3) decrease the rate of overall complications. Aside from several components, or interventions that can vary from institution to institution, these programs share three common modalities: early oral feeding, protocol pain management regimens less dependent on opioid use, and early mobilization (i.e. ambulation). Evidence-based practice has shown that the modalities individually contribute significantly to the program goals except for post-operative ambulation, which has not been shown to increase bowel function although it contributes to decreased pulmonary complications and early discharge of patients. Still, surgeons continue to advocate for early ambulation to aid in the return of bowel function despite the lack of clear evidence supporting this notion.

The investigators propose a randomized, prospective clinical trial exploring the impact that post-operative ambulation has on the outcome of colorectal surgeries, particularly on the return of bowel function and the length of hospital stay. With the use of pedometers to measure physical activity, the investigators will subject patients to either the current traditional post-operative care or one with an aggressive ambulation regimen. Through the use of radiopaque markers, the investigators hope to correlate increased ambulation with increased gastrointestinal motility function to prove the impact of early ambulation on post-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Subject patients are those who will undergo colorectal surgeries at NMCP. Colorectal surgery is defined as any surgery involving the gastrointestinal tract from the ileocecal valve to the dentate line and includes all laparoscopic approaches. This surgery includes, but is not limited to:

  * Ileocecetomy
  * Partial colectomy (including right, left, and sigmoid colectomies)
  * Hartmann procedure
  * Total abdominal colectomy
  * Proctocolectomy
  * Colostomy formation or takedown
  * Low anterior resection
  * Abdominoperineal resection

Exclusion Criteria:

* Reasons for subject exclusion are non-ambulatory conditions are conditions whereby a subject cannot walk or move from place to place. Examples of non-ambulatory conditions include but are not limited to: severe vasculopathy with limiting claudication (leg pain when ambulating due to poor blood flow) of less than 100 meters, all wheelchair bound conditions (anatomically missing both legs without adequate prosthesis, severely limiting pulmonary disease, neurologic disorders - Amyotrophic Lateral Sclerosis, severe multiple sclerosis, paraplegia), fractured leg bones requiring temporary and/or permanent use of a walking aid or any congenital disorders limiting ambulation (osteogenesis imperfecta, muscular dystrophy, cerebral palsy). Any patient who takes Alvimopan (Entereg ®) will be excluded or terminated from the study. Alvimopan is an FDA-approved drug that accelerates bowel motility and is used to prevent and/or treat post-operative ileus. In addition, patients with underlying gastrointestinal motility issues, gastroparesis, chronic constipation, etc or who may have complications who may not be able to ambulate during the hospital course (i.e. prolonged intubated postoperatively) will be excluded as well. Pregnant women will also be excluded from the study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03-31 (Actual); Primary Completion 2014-09-10 (Actual); Study Completion 2014-09-10 (Actual)

PRIMARY OUTCOMES:
Return of bowel function | 1 week
  To demonstrate that increased ambulation as an independent post-operative variable leads to a quicker return of bowel function

SECONDARY OUTCOMES:
Shorter Length of hospitalization | 1 week
  To demonstrate that increased ambulation as an independent post-operative variable leads to a shorter length of hospitalization
Post-operative complications | 30 days
  To demonstrate that increased ambulation as an independent post-operative variable leads to a decrease in the number of overall complications as recorded over a 30-day period post-operatively
Return of normal activities | 30 days
  To demonstrate that increased ambulation as an independent post-operative variable leads to a quicker return of normal activities within a 30-day post-operative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Mentler, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Naval Medical Center Portsmouth, Portsmouth, Virginia, United States